CLINICAL TRIAL: NCT02611791
Title: Radiofrequency Female External Genital Region: a Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1148-8313
Record Dates: First submitted 2015-11-04; First posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Dissatisfaction Appearance of the External Genitalia
Keywords: Treatment by Pulsed Radio Frequency, Collagen, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency (Experimental): Eight RF sessions were performed, with an interval of seven days between them. The application of Radiofrequency in the external genitalia.
  Interventions: Device: Radiofrequency
- Radiofrenquency Off (Sham Comparator): Eight RF sessions were performed, with an interval of seven days between them. The application of Radiofrequency in the external genital which was turned off, but a water-soluble gel was used
  Interventions: Device: Radiofrequency - OFF

INTERVENTIONS:
Device: Radiofrequency — The application of RF was through Tecatherap-VIP unit (VIP-Eletromedicina, Argentina) with bipolar method, using a gauntlet of 2cm, and the coupling electrode, which was located in the sacral region (fig x). For the application, participants were placed in a supine position with legs in lithotomy position, it was used water soluble gel for coupling and slide of the gauntlet. The application in external labia majora was made in the caudal-cranial direction, with constant movement and electrode lightly pressed. (fig) During the session, the heat level was monitored verbally and by infrared digital thermometer. The intensity was gradually increased, and at the time when the temperature reached values between 39-41ºC, the intensity was reduced two points and the procedure was maintained for two minutes.
  Arms: Radiofrequency
Device: Radiofrequency - OFF — The treatment protocol for the control group was identical, differing only in relation to the RF equipment, which was turned off, but a water-soluble gel was used, heated by a resistor, preventing the patient from knowing to which group she belonged. Just the physiotherapist who performed the procedure knew which group the patient belonged to.
  Arms: Radiofrenquency Off

SUMMARY:
OBJECTIVES: The aim of the study is to evaluate the clinical response of the non-ablative radiofrequency (RF) in the outcome cosmetic female external genital and its effect in the sexual function. METHODS: Single blind randomized controlled trial. Sample of 43 women (29 sexual active) with insatisfaction appearance of the external genitalia, 21 (14) in the study group and 22 (15) in the control group. The protocol consisted in 8 sessions of RF once a week. The instruments of evaluation were photo (taken before the first session and eight days after the last session), which were evaluated by the patient and by three health professional (that did not know the group); by the 3 points Likert scale (unsatisfied, unchanged, satisfied) and (worst, unchanged, improved). The sexual function was evaluated by the Female Sexual Function Index (FSFI) before and after, and analyzed by the T Test of Student. The patients' satisfaction and the health professionals' evaluation were analyzed by the chi-squared test and by binomial comparison inter-group and intra-group.

ELIGIBILITY:
Inclusion Criteria:

* were included women aged between 18 and 60 years with unsatisfied the appearance of the external genital, attending the clinical physiotherapy, Bahia, Brazil

Exclusion Criteria:

* Pregnant women, women that were using copper IUD, as well as other with skin lesions in the genital region were excluded from this trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
clinical response | 2 months
  To evaluate the clinical response at radio frequencies of large labia region through the pictures before and after ( assessed by a physiotherapist , gynecologist and dermatologist ).
Patient satisfaction | 2 months
  Patient satisfaction: The response to treatment will be categorized in the absence of improvement; improvement or worsening .

SECONDARY OUTCOMES:
Function Sexual | 2 months
  To evaluate the sexual response after treatment by radio frequency changes in the values of the scores(FSFI) before treatment and at the end.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia V Lordelo, PhD, Principal Investigator — Centro de Atenção ao Assoalho Pélvico - BAHIANA